CLINICAL TRIAL: NCT06358586
Title: Palatability Study of a Novel Paediatric Formulation of Tachipirina® With Strawberry Flavour
Brief Title: New Paediatric Formulation of Tachipirina®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 044(H)MD21176; CRO-PK-21-356 (Other: CRO code)
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: palatability; strawberry flavour; Tachipirina; novel formulation; paediatric
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Intervention Model Description: Single centre, single dose, single-arm, open-label, palatability study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tachipirina® 120 mg/5 mL oral suspension, strawberry flavour (Experimental): All healthy paediatric volunteers administered with the mediation
  Interventions: Drug: Tachipirina® 120 mg/5 mL oral suspension, new flavour

INTERVENTIONS:
Drug: Tachipirina® 120 mg/5 mL oral suspension, new flavour — A single oral dose of the Tachipirina® 120 mg/5 mL oral suspension(10 mL) will be administered to healthy paediatric volunteers under fasting conditions for at least 1 h before IMP administration until completion of palatability assessment.

SUMMARY:
This is a single centre, single dose, single-arm, open-label, palatability study.

The aim of the present study is to investigate the palatability of the newly developed Tachipirina® 120 mg/5 mL oral suspension with strawberry flavour. The study will be conducted in paediatric volunteers that represent the target population for this product.

DETAILED DESCRIPTION:
Twenty (20) healthy paediatric volunteers aged 6-17 years old inclusive will be enrolled in the study.

The primary end-point is to assess the palatability of the new strawberry flavour after single dose administration of the Investigation Medicine Product (IMP) through a questionnaire.

The secondary end-points is to monitor the safety and tolerability data after single dose administration of the Investigation Medicine Product (IMP).

ELIGIBILITY:
Inclusion Criteria:

* Sex and Age: males or females, 6-17 years old inclusive
* Body Mass Index: males/females not classified as overweight based on the applicable body mass index chart for sex and age
* Informed consent and assent: signed written informed consent by both parents/legal representatives unless only one has legal authority. Signed written informed assent for 14-17 years old inclusive adolescents or written informed assent for 11-13 years old inclusive children or oral informed assent for 6-10 years old inclusive children.
* Full comprehension: ability of the paediatric volunteer and parent(s)/legal representative(s) to comprehend the full nature and purpose of the study, including possible risks and side effects; ability of the paediatric volunteer and parent(s)/legal representative(s) to co-operate with the Investigator and to comply with the requirements of the entire study
* Ascertained tolerability to paracetamol: history of intake of Tachipirina® or its active ingredient, i.e., paracetamol, with no consequent adverse reaction

Exclusion Criteria:

* Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
* Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Diseases: history of significant renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; mouth lesions or any other oral mucosa alteration that may interfere with the aim of the study according to the Investigator's opinion
* Medications: medications, including over the counter medications and herbal remedies for 2 weeks before the start of the study that may interfere with the aim of the study according to the Investigator's opinion. Hormonal contraceptives for child-bearing potential females (i.e., post-menarche) will be allowed
* Tobacco: smokers will not be admitted
* Investigative drug studies: participation in the evaluation of any investigational medicinal product for 3 months before this study. The 3-month interval will be calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
* Diet: abnormal diets or substantial changes in eating habits in the 4 weeks before this study that may interfere with the aim of the study according to the Investigator's opinion
* SARS-CoV-2 test: positive Covid-19 Antigen Rapid Test at screening of paediatric volunteer or parent(s)/legal representative(s)
* Drug test: only for adolescents 12-17 years old inclusive, positive drug test at screening
* Alcohol breath test: only for adolescents 12-17 years old inclusive, positive alcohol breath test at screening
* Pregnancy: only for child-bearing potential females (i.e., post-menarche), positive or missing pregnancy test at screening

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-04-09 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Palatability of new flavour - Taste (1) | 15 minutes after investigational medicinal product administration
  Subject are asked: How do you describe the taste of this medication? The corresponding answer are sweet, salty, sour, bitter.
Palatability of new flavour - Taste (2) | 15 minutes after investigational medicinal product administration
  Subject are asked: How much do you like the taste of this medication? The corresponding answer are given using a hedonic facial scale i.e. the 7-points rating Chen scale in which descriptive replies are associated to images showing different facial expressions to allow the children to easily quantitate their sensory experiences. For the Chen scale, a numeric score will be assigned by the Investigator as follows:
  * Very bad = 1
  * Bad = 2
  * Just a little bad = 3
  * Not sure = 4
  * Just a little good = 5
  * Good = 6
  * Very good = 7
Palatability of new flavour - Smell | 15 minutes after investigational medicinal product administration
  Subject are asked: How much do you like the smell of this medication? The corresponding answer are given using a hedonic facial scale i.e. the 7-points rating Chen scale in which descriptive replies are associated to images showing different facial expressions to allow the children to easily quantitate their sensory experiences. For the Chen scale, a numeric score will be assigned by the Investigator as follows:
  * Very bad = 1
  * Bad = 2
  * Just a little bad = 3
  * Not sure = 4
  * Just a little good = 5
  * Good = 6
  * Very good = 7
Palatability of new flavour - Aftertaste (1) | 15 minutes after investigational medicinal product administration
  Subject are asked: Do you feel an aftertaste after the administration of this medication? The corresponding answer are Yes or No.
Palatability of new flavour - Aftertaste (2) | 15 minutes after investigational medicinal product administration
  If Subjects reply Yes to the previous question they are asked: Do you describe the aftertaste of this medication? The corresponding answer are sweet, salty, sour, bitter.
Palatability of new flavour - Aftertaste (3) | 15 minutes after investigational medicinal product administration
  If Subjects replies Yes to the previous question they are asked: How much do you like the aftertaste of this medication? The corresponding answer are given using a hedonic facial scale i.e. the 7-points rating Chen scale in which descriptive replies are associated to images showing different facial expressions to allow the children to easily quantitate their sensory experiences. For the Chen scale, a numeric score will be assigned by the Investigator as follows:
  * Very bad = 1
  * Bad = 2
  * Just a little bad = 3
  * Not sure = 4
  * Just a little good = 5
  * Good = 6
  * Very good = 7
Palatability of new flavour - Texture (mouthfeel) | 15 minutes after investigational medicinal product administration
  Subject are asked: How do you describe the texture of this medication in the mouth? The corresponding answer are Thin, thick, gritty.
Palatability of new flavour - Overall | 15 minutes after investigational medicinal product administration
  Subject are asked: In general, how much do you like this medication?The corresponding answer are given using a hedonic facial scale i.e. the 7-points rating Chen scale in which descriptive replies are associated to images showing different facial expressions to allow the children to easily quantitate their sensory experiences. For the Chen scale, a numeric score will be assigned by the Investigator as follows:
  * Very bad = 1
  * Bad = 2
  * Just a little bad = 3
  * Not sure = 4
  * Just a little good = 5
  * Good = 6
  * Very good = 7

SECONDARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | Through study completion, an average of 2 weeks.
  Number of TEAEs after single dose administration of the investigational medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, Principal Investigator — CROSS Research S.A. - Phase I Unit,
Locations (1):
- CROSS Research S.A. - Phase I Unit,, Arzo, Switzerland